CLINICAL TRIAL: NCT03505463
Title: The Neuroinflammatory Response and Biomarkers in Acute Traumatic Spinal Cord Injury: A Pilot Study
Brief Title: The Neuroinflammatory Response and Biomarkers in Acute Traumatic Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Spinal Cord Injury Centre of Western Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 490-13-3632
Record Dates: First submitted 2018-04-11; First posted 2018-04-23 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injury, Acute
Keywords: Spinal cord injury; Biomarkers; Inflammation; Trauma
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation; Wounds and Injuries | interventions — Blood Specimen Collection; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Injured participants
  Interventions: Other: Blood samples; Other: Cerebrospinal fluid sample; Other: Clinical examination
- Healthy participants
  Interventions: Other: Blood samples; Other: Cerebrospinal fluid sample

INTERVENTIONS:
Other: Blood samples — Three blood samples will be collected from the injured participants. The assessment points are <72 hours, 7 days and 365 days post-injury.
  One blood sample will be collected from the healthy participants. The collection will be performed as part of clinical diagnostic at the Department of Neurology at Aarhus University Hospital.
  Laboratory analysis of the collected samples comprise Flow Cytometry and assay techniques.
Other: Cerebrospinal fluid sample — Three cerebrospinal fluid samples will be collected from the injured participants. The assessment points are <72 hours, 7 days and 365 days post-injury.
  The collected samples will be analysed by Flow Cytometry and assay techniques. One cerebrospinal fluid sample will be collected from the healthy participants. The collection will be performed as part of clinical diagnostic at the Department of Neurology at Aarhus University Hospital.
  Laboratory analysis of the collected samples comprise Flow Cytometry and assay techniques.
Other: Clinical examination — Clinical examinations will be performed at <72 hours, 7 days and 365 days post-injury.
  Groups: Injured participants

SUMMARY:
The study is a prospective cohort study designed to assess the diagnostic and prognostic potential of biomarker measurement in acute traumatic spinal cord injury (TSCI), and to examine the neuroinflammatory response to acute TSCI.

DETAILED DESCRIPTION:
TSCI is an incurable condition with devastating consequences. The physical, psychosocial and financial implications in addition to a variable recovery and an uncertain prognosis have a profound impact on quality of life.The pathophysiology of TSCI is dual consisting of a primary injury and a secondary injury. The immediate trauma to the spinal cord and nerve roots causes the primary injury, while a prolonged cascade of events causes the secondary injury. The neuroinflammatory response is considered to be an important event. Current clinical measures to evaluate acute TSCI consist of clinical examination and routine imaging modalities. These measurements are inaccurate to assess injury severity, prognosis, and therapeutic efficacy, especially in the early acute phase. Biomarker measurement may provide a more accurate measure.

This study aim to assess the diagnostic and prognostic potential of biomarker measurement in acute TSCI, and to examine the neuroinflammatory response to acute TSCI. To achieve this, immune cells, cytokines, autoantibodies and structural proteins will be analysed in blood and cerebrospinal fluid by Flow Cytometry and assay techniques. These analyses will be correlated to clinical outcome assessed according to international standards.

Hopefully, this will contribute with new knowledge of the neuroinflammatory response and biomarkers in acute TSCI, and provide the needed knowledge for conducting futures trials in novel therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury (Bony level C1-L1)
* ISNCSCI score A-C upon inclusion.
* Age >18-70 years.

Exclusion Criteria:

* Prior major spine surgery in the traumatised location.
* Major co-morbidities or co-injuries.
* Penetrating spinal cord injury.
* >72 hours from injury to sample collection.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consist of 10 acute traumatic spinal cord injured participants admitted to the Department of Neurosurgery at Aarhus University Hospital and 20 healthy participants investigated at the Department of Neurology at Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | <72 hours, 7 days and 365 days post-injury.

SECONDARY OUTCOMES:
Walking Index for Spinal Cord Injury II (WISCI II) | 365 days post-injury
The Spinal Cord Independence Measure III (SCIM III) | 365 days post-injury
Visual Analogue Pain Score (VAS) | 365 days post-injury
  VAS will be used to assess pain intensity. VAS is a scale ranging from 0 to 10 where "No pain" gives a score of 0 and "worst imaginable pain" gives a score of 10.
International Spinal Cord Injury Dataset for core | 365 days post-injury
International Spinal Cord Injury Dataset for pain | 365 days post-injury
International Spinal Cord Injury Dataset for bladder | 365 days post-injury
International Spinal Cord Injury Dataset for bowel | 365 days post-injury
International Spinal Cord Injury Dataset for sexual function | 365 days post-injury

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wichmann TO, Kasch H, Dyrskog S, Hoy K, Moller BK, Krog J, Hoffmann HJ, Hviid CVB, Rasmussen MM. Glial fibrillary acidic protein is a robust biomarker in cerebrospinal fluid and peripheral blood after traumatic spinal cord injury: a prospective pilot study. Acta Neurochir (Wien). 2023 Jun;165(6):1417-1425. doi: 10.1007/s00701-023-05520-x. Epub 2023 Feb 15. PMID 36790588